CLINICAL TRIAL: NCT04932083
Title: Intrathecal Midazolam is a Comparable Alternative to Fentanyl and Nalbuphine as Adjuvant to Bupivacaine in Spinal Anesthesia for Elective Cesarean Section; a Randomized Controlled Double-blind Trial
Brief Title: Intrathecal Midazolam, Fentanyl and Nalbuphine as Adjuvants to Bupivacaine in Spinal Anesthesia for Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Samar Rafik Mohamed Amin, lecturer of anesthesia and surgical ICU, Benha University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RC6-5-2021
Record Dates: First submitted 2021-06-14; First posted 2021-06-18 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain | interventions — Bupivacaine; Fentanyl; Nalbuphine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Bupivacaine (Placebo Comparator): patients will receive 2.5 ml of 0.5% hyperbaric bupivacaine (12.5 mg) plus 0.5 ml sterile water.
  Interventions: Drug: Bupivacaine
- Fentanyl (Experimental): patients will receive 2.5 ml of 0.5% hyperbaric bupivacaine (12.5 mg) plus 0.5 ml fentanyl (25µg).
  Interventions: Drug: Fentanyl
- Nalbuphine (Experimental): patients will receive 2.5 ml of 0.5% hyperbaric bupivacaine (12.5 mg) plus 0.8 mg nalbuphine hydrochloride in 0.5 ml sterile water.
  Interventions: Drug: Nalbuphine
- Midazolam (Experimental): patients will receive 2.5 ml of 0.5% hyperbaric bupivacaine (12.5 mg) plus 2mg of midazolam in 0.5 ml sterile water.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Bupivacaine — patients will be put in the sitting position and lean forward. After sterilization, Dural puncture will be performed at L4-L5 interspace or L3-L4 with a 25 gauge Quincke spinal needle.
  patients will receive the local anesthetic dose of 0.5% heavy bupivacaine (12.5 mg) and 0.5 ml of sterile water will be added.
  Arms: Bupivacaine
Drug: Fentanyl — patients will be put in the sitting position and lean forward. After sterilization, Dural puncture will be performed at L4-L5 interspace or L3-L4 with a 25 gauge Quincke spinal needle.
  patients will receive the local anesthetic dose of 0.5% heavy bupivacaine (12.5 mg) and 0.5 ml of fentanyl (25µg) will be added.
  Arms: Fentanyl
Drug: Nalbuphine — patients will be put in the sitting position and lean forward. After sterilization, Dural puncture will be performed at L4-L5 interspace or L3-L4 with a 25 gauge Quincke spinal needle.
  patients will receive the local anesthetic dose of 0.5% heavy bupivacaine (12.5 mg) and 0.8 mg nalbuphine hydrochloride in 0.5 ml sterile water will be added.
  Arms: Nalbuphine
Drug: Midazolam — patients will be put in the sitting position and lean forward. After sterilization, Dural puncture will be performed at L4-L5 interspace or L3-L4 with a 25 gauge Quincke spinal needle.
  patients will receive the local anesthetic dose of 0.5% heavy bupivacaine (12.5 mg) and 0.4 ml of midazolam (2mg) + 0.1 ml of sterile water will be added.
  Arms: Midazolam

SUMMARY:
The main limitations of spinal anesthesia are its short duration of action and do not provide prolonged postoperative analgesia when it is performed only with local anesthetics. Adding adjuvants drugs to intrathecal local anesthetics improves quality and duration of spinal blockade, and prolongs postoperative analgesia. It is also possible to reduce dose of local anesthetics, as well as total amount of systemic postoperative analgesics.

DETAILED DESCRIPTION:
Several spinal adjuvants have been used to improve spinal anesthesia quality and to prolong postsurgical analgesia; Intrathecal opioids are the most commonly utilized. Intrathecal opioids cause analgesia by binding to opioid receptors in the dorsal horn of the spinal cord. They prolong the duration of analgesia and allow early ambulation of patients.

Fentanyl, a short-acting lipophilic opioid, is known to augment the quality of subarachnoid block in many studies. However, worrisome adverse effects such as pruritus, urinary retention, post-operative vomiting, and respiratory depression limit the use of opioids.

Nalbuphine is a synthetic opioid with mixed agonist antagonist effect. It binds to both mu- and kappa receptors; binding of nalbuphine to mu receptors competitively displaces other mu-agonists from these receptors without any agonist activity, therefore decreasing the side effects on mu agonist (nausea, vomiting, respiratory depression, urinary retention, pruritis, and prolonged sedation). While when binding to kappa receptors, nalbuphine has agonist effect (analgesic effect) through the kappa receptors distributed in the brain and spinal cord. There have been no documented studies of nalbuphine neurotoxicity.

Midazolam is a short acting benzodiazepine with anxiolytic, sedative, anticonvulsant and muscle relaxant effects, influencing GABA receptor and influence on neurons by entering chloride into them. It is water soluble in its acid formulation but is highly lipid soluble in vivo. It has been reported to have a spinally mediated anti-nociceptive effect. Previous studies have shown that intrathecal administration of midazolam added to bupivacaine improves the duration and quality of spinal anesthesia.

This study is carried out to evaluate and compare the effects of intrathecal midazolam (2 mg), fentanyl (25 micrograms) and nalbuphine (800 micrograms) as additives to intrathecal hyperbaric bupivacaine (0.5 %) with regards to: onset and duration of sensory block, onset and duration of motor block, duration of effective analgesia postoperative, side effects associated with the drug.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status I and ASA II
2. Age from 18-40 years
3. Scheduled to undergo elective cesarean section under spinal anesthesia.

Exclusion Criteria:

1. ASA physical status III or IV patients.
2. Patients refuse spinal anesthesia.
3. Patients physically dependent on narcotics or benzodiazepine.
4. Patients with history of drug allergy to one of used adjuvants.
5. Patients with gross spinal abnormality, localized skin sepsis, hemorrhagic diathesis or neurological involvement/ diseases and any contraindication for spine.
6. Patients who are unable to communicate.
7. Morbid obesity.
8. Failure of spinal blockade.
9. Complicated pregnancy.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — full term parturients undergo elective cesarean section,
Enrollment: 100 (Actual)
Dates: Start 2021-06-20 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-02-24 (Actual)

PRIMARY OUTCOMES:
Duration of effective analgesia | 24 hours postoperative
  it is the time interval from the subarachnoid block to the first analgesic intervention (VAS >3)

SECONDARY OUTCOMES:
The onset of sensory block: | 2 minutes for ten minutes, every 5 minutes for the next 20 minutes after intrathecal injection
  it is the time from end of intrathecal injection to absence of pain at T5 dermatome.
Duration of complete sensory block: | 12 hours postoperative
  it is the time interval from the subarachnoid block to the first sensation of pain (VAS >0).
Onset of complete motor blockade | every 2 minutes for 10 minutes after intrathecal injection
  it is the time per minutes from intrathecal injection until Bromage scale to be 3.
Duration of motor block: | 6 hours postoperative
  it is the time per minutes from intrathecal injection until Bromage score 0.
Total dose of analgesic consumption | 24 hours postoperative
  if VAS pain score >3, intravenous 30 mg keterolac will be administered and can be repeated after 6 h if needed. If the mother was still complaining of pain or the VAS is still greater than 3 after 20 min from ketorolac injection, she will be given intravenous pethidine in a dose of 0.5 mg/kg.
Maternal adverse effects | 24 hours postoperative
  All mothers will be monitored for the associated adverse effects such as postoperative nausea and vomiting (PONV), sedation, pruritus, hypotension, bradycardia, shivering, and respiratory depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Samar Rafik Amin, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No